CLINICAL TRIAL: NCT02900001
Title: Routinely Deferred Versus Early Invasive Strategy in Chinese Patients of 75 Years or Older With Non-ST-elevation Myocardial Infarction - a Multicenter, Open-label, Randomized Controlled Clinical Trial.
Brief Title: Routinely Deferred Versus Early Intervention in Elderly Patients With Non-ST-elevation Myocardial Infarction
Acronym: DEAR-OLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Yuejin Yang, vice president of Fuwai Hospital, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LHJJ201510626
Record Dates: First submitted 2016-08-24; First posted 2016-09-14 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-09

CONDITIONS: Non-ST Elevation Myocardial Infarction
Keywords: myocardial infarction; invasive strategy; elderly; deferred
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early invasive strategy (Active Comparator): Patients undergo coronary angiography within 24 hours after admission and have percutaneous coronary intervention or coronary artery bypass grafting as soon as possible during the index hospitalization if appropriate.
  Interventions: Procedure: early coronary angiography
- Deferred invasive strategy (Experimental): Patients undergo coronary angiography and appropriate revascularization after at lest 72 hours from admission in the index hospitalization.
  Interventions: Procedure: delayed coronary angiography

INTERVENTIONS:
Procedure: early coronary angiography — Routine coronary angiography and revascularization if appropriate within 24 hours
  Arms: Early invasive strategy
Procedure: delayed coronary angiography — Routine coronary angiography and revascularization if appropriate after 72 hours
  Arms: Deferred invasive strategy

SUMMARY:
This study is to evaluate the efficacy and safety of a routinely deferred invasive strategy in comparison with an early invasive strategy in Chinese elderly patients of 75 years or older with non-ST elevation myocardial infarction, aiming to test the hypothesis that routinely deferred invasive strategy is not inferior to early invasive strategy in such an elderly group of patients.

DETAILED DESCRIPTION:
This study aims to enroll 696 elderly patients with non-ST elevation myocardial infarction (NSTEMI) from 20 hospitals throughout mainland China.. Consective patients of 75 years or older with a diagnosis of NSTEMI will be suitable for enrollment. Written informed consent form will be obtained from every patients. Initially stabilized patients with an ischemic episode within 24 hours before admission will be randomized and others will be registered. For randomization, the patients' brief information will be entered in a central randomization system to generate a random number.

According to the random number, each patient will be randomly assigned to early invasive therapy versus routinely deferred invasive strategy. All patients will initiate dual antiplatelet therapy (aspirin+P2Y12 inhibitor) and continued till the end of follow-up at one year. For patients assigned to early invasive group, a loading dose of antiplatelet agent should be given, unless contraindicated. Anticoagulation, anti-ischemic agents, statin and other guideline recommended medicine will be given according to physician in charge according to guideline.

Patients assigned to early invasive strategy will undergo coronary angiography within 24 hours after admission and have percutaneous coronary intervention or coronary artery bypass grafting as soon as possible during the index hospitalization if appropriate. Patients assigned to deferred invasive strategy will undergo coronary angiography and subsequent revascularization after at lest 72 hours after admission and in the index hospitalization. Patients who undergo percutaneous coronary intervention can receive a glycoprotein IIb/IIIa inhibitor if indicated and upfront use of glycoprotein IIb/IIIa inhibitors is discouraged. The choice of intervention or surgery and the choice of complete or staged revascularization will be determined by the operator according to coronary anatomy and consistent with current practice guidelines. Patients assigned to deferred strategy should undergo urgent coronary angiography and revascularization accordingly if indicated during the period of time waiting for catheterization. Such procedure will be adjudicated as an endpoint. Elective percutaneous coronary intervention on non-culprit vessels, in either study arm, can take place sometime after the index procedure with the goal to achieve complete revascularization. Such staged procedures will not be deemed as an adverse event.

Specific data for acquisition:

Research demographics: age, height, weight, body mass index, medications at randomization, pertinent medical/family/social history, i.e., hypertension, hypercholesterolemia, diabetes mellitus, current tobacco use, history of prior myocardial infarction, PCI or CABG. This data will be gathered by research coordinator through interviewing patient and checking patient's medical record.

Procedural: Exact time of onset of ischemic symptoms, of admission, of randomization, and of undertake coronary angiography will be noted by a supplemental chart, along with important information like the evidence of occurrence of an endpoint. Blood concentration of hemoglobin, BNP/NT-proBNP, creatinine, cardiac troponin and C-reaction protein will be tested at admission. First electrocardiography and echocardiography will be recorded. Thrombolysis In Myocardial Infarction flow will be recorded before and after PCI procedure, and the images will be copied to calculate the SYNTAX score afterwards.

After hospital discharge, the research coordinator will contact the patient at specified intervals （30 days after discharge, 180 days and 365 days after randomization） to determine if an endpoint has been met.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 75 years or older
2. Elevated cardiac troponin;
3. Ischemic symptom or ST-segment depression in ECG；
4. Newly onset of myocardial ischemia within 24 hours;
5. Written Informed Consent obtained.

Exclusion Criteria:

1. Type 2 MI (secondary to tachyarrhythmias, uncontrolled hypertension, anemia, hyperthyroidism, acute pulmonary infection, or fever)
2. Secondary elevation of cardiac troponin (e.g. renal insufficiency, heart failure, et al.)
3. Persistent ST-segment elevation or new pathologic Q wave indicating STEMI
4. Ongoing myocardial ischemia despite intensive medical treatment after admission
5. Refractory acute heart failure that can not be well controlled despite treatment for 24 hours
6. Hemodynamic instability or cardiac shock on admission
7. History of cardiac arrest or ventricular tachycardia/fibrillation after symptom onset
8. Concomitant use of oral anticoagulants for atrial fibrillation or thromboembolism diseases
9. PCI or bypass surgery within 30 days before randomization
10. History of contrast agent allergy
11. Baseline serum creatinine of >2.5 mg/dl or calculated creatinine clearance rate of <30 ml/min
12. Known bleeding diathesis or contraindications to dual antiplatelet treatment like active internal bleeding
13. Gastrointestinal and genitourinary bleeding of clinical significance within 6 weeks before randomization
14. History of stroke within 3 months
15. infectious diseases or fever
16. Life expectancy < 6 months

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 696 (Estimated)
Dates: Start 2016-12-01 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2019-10-30 (Estimated)

PRIMARY OUTCOMES:
Composite endpoint of all-cause mortality, non-lethal myocardial infarction, stroke and urgent revascularization | 1 year

SECONDARY OUTCOMES:
No reflow | during PCI
  composite and Individual component
All-cause mortality | 30 days after discharge, 6 months and 1 year after randomization
  composite and Individual component
Non-lethal myocardial infarction | 30 days after discharge, 6 months and 1 year after randomization
  composite and Individual component
Severe recurrent ischemia | 30 days after discharge, 6 months and 1 year after randomization
  composite and Individual component
Stroke | 30 days after discharge, 6 months and 1 year after randomization
  composite and Individual component
Major bleeding | 30 days after discharge, 6 months and 1 year after randomization
  composite and Individual component

CONTACTS AND LOCATIONS:
Overall Officials: Yuejin Yang, M.D., PhD., Principal Investigator — National Center for Cardiovascular Diseases, Chinese Academy of Medical Sciences and Peking Union Medical College, Fuwai Hospital
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leng WX, Yang J, Li W, Wang Y, Yang YJ; DEAR-OLD investigators. Rationale and design of the DEAR-OLD trial: Randomized evaluation of routinely Deferred versus EARly invasive strategy in elderly patients of 75 years or OLDer with non-ST-elevation myocardial infarction. Am Heart J. 2018 Feb;196:65-73. doi: 10.1016/j.ahj.2017.10.022. Epub 2017 Nov 5. PMID 29421016